CLINICAL TRIAL: NCT03130387
Title: Prevalence of Cesarean Section Niche in Women With Unexplained Abnormal Uterine Bleeding
Acronym: Niche
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Head of Early Cancer Detection Unit, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEldawa
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Cesarean Section; Dehiscence; Abnormal Uterine Bleeding
Keywords: Hytsteroscopy
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Intervention Model Description: Hysteroscopic examination for patients with AUB
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Office hysteroscopy (Other): Examinatin with Office hysteroscope for women with abnormal uterine bleeding who had a history of previous cesarean section
  Interventions: Device: Office Hysteroscope

INTERVENTIONS:
Device: Office Hysteroscope — Diagnosis of C.S niche in patients wit AUB by office hysteroscope

SUMMARY:
Prevalence of Cesarean Section Niche in women With Unexplained Abnormal Uterine Bleeding

DETAILED DESCRIPTION:
Prevalence of Cesarean Section Niche as diagnosed by office hysteroscopy and transvaginal sonography in women With Unexplained Abnormal Uterine Bleeding

ELIGIBILITY:
Inclusion Criteria:

Patients with a history of cesarean section who are complaining of abnormal uterine bleeding with the following criteria :

* Normal complete blood count apart from paramaters of anemia
* Not using drugs affecting coagulation profile
* Bleeding is not related to pregnancy
* Not using intrauterine contraceptive devices or hormonal contraceptives
* By ultrasonography : no abnormalities in the pelvis e.g benign or malignant tumors , ovarian cysts or tumors
* No evidence of cervical abnormalities as cause of bleeding with cervical examination or cervical smears

Exclusion Criteria:

* Any patient not fulfilling the inclusion criteria
* If the patient refused the technique ( office hysteroscopy )

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females only
Enrollment: 95 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of cisarean section niche | 1 year
  Prevalence of cisarean section niche in women complainig of unexplained abnormal uterine bleeding

IPD SHARING:
Plan to Share IPD: Undecided